CLINICAL TRIAL: NCT05321342
Title: Coaching Late Elementary School Teachers in Bullying Detection and Intervention (Bullying Classroom Check-Up)
Brief Title: Coaching Teachers in Bullying Detection and Intervention
Acronym: BCCU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Virginia (Other); Sheppard Pratt Health System (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD102491-01A1 (NIH); 20-018301 (Other: Children's Hospital of Philadelphia); IRB00015114 (Other: Johns Hopkins Bloomberg School of Public Health)
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Intervention; Control
Keywords: Bullying; Aggression; Classroom Climate; Teacher Coaching; Simulation
MeSH Terms: conditions — Bullying; Aggression

STUDY DESIGN:
Intervention Model Description: Half of the schools each year will be recruited from the School District of Philadelphia (SDP) and half from the Anne Arundel County Public Schools (AACPS) in Maryland. Within site, half of the schools will be assigned to the BCCU intervention and half will be in the control ("business as usual" condition; data collection only, plus an offer of a classroom management PD after research participation ends).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will receive Professional Development and Coaching (CCU)
  Interventions: Behavioral: Bullying Classroom Check-Up (BCCU)
- Control group (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Bullying Classroom Check-Up (BCCU) — BCCU professional development (PD) modules will be provided to all staff in intervention schools as part of their standard, school-approved professional development practices to provide knowledge and awareness for bullying identification, prevention, and intervention. In addition, consented 3rd-5th grade teachers will participate in the BCCU intervention. The coaching follows the original Classroom Check-Up model (Reinke, Herman, & Sprick, 2011), embedding 5 steps (i.e., assessment of the classroom, feedback to teacher, goal setting and plan, ongoing coaching and guided practice in the TeachLivE© mixed-reality simulator [developed at the University of Central Florida (UCF); Dieker, Hynes, Hughes, & Smith, 2008], and self-monitoring) and utilizing motivational interviewing (Miller & Rollnick, 2012) to empower teacher practice change.
  Arms: Intervention group

SUMMARY:
The investigators' overall objective is to demonstrate the efficacy of the Bullying Classroom Check-Up (BCCU) on elementary aged students' aggressive and bullying behaviors, teacher practices, and student and teacher relationships. The investigators' principal hypothesis is that the BCCU will improve students' aggression and bullying behaviors and their perceptions of the school climate and relationships in the building as well as teacher practices.

DETAILED DESCRIPTION:
Aim 1: Examine the Efficacy of the Bullying Classroom Check-Up (BCCU) at improving child aggressive and bullying behaviors For this aim, the study team will examine student self-report measures and classroom observational data at post-test (end of year 1) and in the follow-up assessment (winter of following school year). The study team will focus on their own aggression and bullying behavior as well as their perceptions of the general bullying climate, rating of safety, and positive bystander behaviors (i.e., how students respond to bullying when they witness it). The study team hypothesize that children in schools randomized to the BCCU condition will be less likely to engage in aggression and bullying, will rate the general bullying climate (i.e., perceptions that bullying is a problem and that adults/students do enough to stop bullying) and sense of safety more positively, and engage in more positive bystander behaviors than children in schools randomized to the control condition.

Aim 2: Examine the efficacy of the BCCU at improving teacher practices and relationships For this aim, the study team will examine teacher and aggregated student self-report measures and classroom observational data at post-test (end of year 1) and in the follow-up assessment (winter of following school year). The study team will focus on teacher self-reported, observed, and student-reported classroom practices as well as perceptions from teachers and students about relationships within the school. The investigators' hypotheses are that teachers in the BCCU condition will engage in more preventive classroom management and intervention strategies (e.g., modeling social emotional competencies such as empathy) in response to bullying than teachers in the control condition, and that teacher-student and student-student relationships will be more positive in classrooms in the BCCU condition than in the control condition.

Exploratory Aim 3: Explore the moderating role of fidelity in the main outcomes of interest. Explore the mediating role of teacher self-efficacy and behavior management practices on distal outcomes.

For this exploratory aim, the study team will examine how fidelity indicators (e.g., dosage, coach adherence, as reported by coaches) moderates intermediate teacher outcomes (e.g., teacher practices) within the main effect models. The study team will also examine how changes in teacher intermediate outcomes (e.g., teacher efficacy and practices) relate to the follow-up year's classroom climate (e.g., relationships) as reported by students (aggregated) and teachers in mediation models.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Schools 32 schools will be selected based on the following inclusion criteria:

1. Urban to urban fringe districts in the Northeast US
2. Predominately minority student body (> 65%)
3. Relatively large school with at least two 3rd, 4th, and 5th grade classrooms

Inclusion Criteria - Teachers 1) Teachers of 3rd-5th grade regular education classrooms employed by the participating school sites who provide their consent for participation.

Inclusion Criteria - Students

1) All students of consented teachers will be eligible to participate in survey activities.

Exclusion Criteria:

Exclusion Criteria - Teachers

1. Teachers in grades other than 3, 4, or 5 during the first year
2. Special education teachers
3. Specials (e.g., art, music) teachers

Exclusion Criteria - Students

1. Students who do not speak English.
2. Special education students who are not integrated within the regular education classroom (i.e., receive education in self-contained classrooms).

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Teacher Prevention/Intervention Strategies | Administered at baseline (before the intervention is launched)
  As self-reported by both teacher and students 'handling of aggression and bullying' designed for this study as well as an observational measure, the ASSIST of proactive behavior management for prevention.
Safety and aggression climate | Administered at baseline (before the intervention is launched)
  As self-reported by both teacher and students on surveys using the Maryland Safe and Supportive Schools (MDS3) School Climate scales on safety, rules and consequences, and the general aggression/bullying climate as well as an observational measure, the ASSIST of the disruptive behaviors in the classroom.

SECONDARY OUTCOMES:
Teacher use of social emotional learning (SEL) | 3 classroom observations at baseline (before the intervention is launched)
  Collected by research team-hired observers trained in an observational measure, called the ASSIST, assessing use of SEL in the classroom 3 classroom observations at baseline.
Bullying and Positive Bystander Behaviors | Administered at baseline (before the intervention is launched)
  As self-reported by both teacher and students on surveys using the MDS3 School Climate scales on experiences as a victim of bullying, bystander responses as well as an observational measure, the ASSIST of the aggressive behaviors in the classroom
Teacher Efficacy and burnout | Administered at baseline (before the intervention is launched)
  As self-reported by teacher using a measure of emotional exhaustion/burnout and behavior management self-efficacy
Teacher and student connectedness | Given first at baseline (before the intervention is launched)
  As self-reported by both teacher and students on surveys using the MDS3 School Climate scales on teacher connectedness and student connectedness (teacher version) and student-teacher and student-student relationships (student version)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Pas, PhD, Principal Investigator — Johns Hopkins University; Tracy Waasdorp, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No